CLINICAL TRIAL: NCT04114097
Title: The Effects of Topical Corticosteroid Use on Insulin Sensitivity and Bone Turnover
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jacob Thyssen (Other)
Collaborators: LEO Pharma (Industry)
Responsible Party: Sponsor-Investigator, Jacob Thyssen, Professor, consultant, University Hospital, Gentofte, Copenhagen
Organization: University Hospital, Gentofte, Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: H-18064175
Record Dates: First submitted 2019-10-01; First posted 2019-10-03 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Atopic Dermatitis; Atopic Eczema
Keywords: topical corticosteroids; topical calcineurin inhibitors
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Betamethasone Valerate; Tacrolimus

STUDY DESIGN:
Intervention Model Description: randomised, two-arm, active comparator, double-dummy, double-blinded trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Betamethasone-17-valerat + placebo ointment (Experimental): Atopic dermatitis patients: topical treatment with twice daily full-body ointment containing corticosteroid ("Betnovate", betamethasone dipropionate ointment 0.1%) and placebo
  Interventions: Drug: Betnovate, betamethasone dipropionate ointment 0.1% and placebo
- Tacrolimus ointment (Active Comparator): Atopic dermatitis patients: topical treatment with twice daily full-body ointment containing calcineurin inhibitor ("Protopic", tacrolimus ointment 0.1%)
  Interventions: Drug: Protopic, tacrolimus ointment 0.1%

INTERVENTIONS:
Drug: Betnovate, betamethasone dipropionate ointment 0.1% and placebo — Explore the systemic effects of Betnovate
  Arms: Betamethasone-17-valerat + placebo ointment
Drug: Protopic, tacrolimus ointment 0.1% — Compare the systemic effects of Betnovate to Protopic
  Arms: Tacrolimus ointment

SUMMARY:
The investigators believe that the emerging epidemiological evidence connecting topical use of corticosteroids to the development of type 2 diabetes and osteoporosis point to potentially massive, yet clinically unacknowledged problems associated with topical corticosteroid treatment. Using state-of-the-art methodology, the present study will delineate the impact of topical corticosteroid use on insulin sensitivity and bone turnover markers in patients with atopic dermatitis and, thus, provide important data that may have implications for millions of people using topical corticosteroids.

ELIGIBILITY:
Inclusion criteria

* Age 18-75 years
* AD according to the Hanifin and Rajka Criteria24
* AD for at least 3 years
* BMI ≤ 30 kg/m2
* Haemoglobin A1c (HbA1c) ≤ 42 mmol/mol (6.0%)
* Normal haemoglobin (men: 8.3-10.5 mmol/L and women 7.3-9.5 mmol/L. A 5% deviation will be allowed if the patient besides this is healthy)
* Informed consent
* In general patients should not be diagnosed with diseases that may affect or be affected by the study/treatment (evaluated by a doctor) (such as untreated skin infections, acne vulgaris (beside face region), a skin barrier defect, such as Netherton's syndrome, lamellar ichthyosis, generalized erythroderma or cutaneous Graft Versus Host Disease, congenital or acquired immunodeficiencies or in patients on therapy that cause immunosuppression, and Protopic ointment should not be applied to lesions that are considered to be potentially malignant or pre-malignant. Further patients should not suffer from kidney or liver disease/insufficiency. See the SPC for Protopic and Betnovate.)

Exclusion criteria

* Diagnosed diabetes mellitus
* Other chronic inflammatory diseases (including but not limited to rheumatoid arthritis, inflammatory bowel disease etc) beside AD and non-treatment demanding rhinitis or asthma (treated within the last 4 weeks)
* Pregnancy (a urine test will be done at every visit and birth control is required, see below*)
* Breast feeding
* Treatment with drugs that might affect the glucose metabolism beside TCS within a month prior to the project
* Daily smoker, alcoholic, or drug abuser
* Hypersensitivity to Protopic or Betnovate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Change in whole-body insulin sensitivity | Baseline, after 14 days daily treatment, and after 4 weeks of twice daily treatment twice weekly
  Change in whole-body insulin sensitivity during treatment with topical corticosteroid use compared to the control group treated with topical calcineurin inhibitors. Insulin sensitivity will be assessed by the hyperinsulinaemic euglycaemic clamp method with glucose and glycerol tracer and indirect calorimetry (rate of disappearance (Rd)).

CONTACTS AND LOCATIONS:
Overall Officials: Jacob P Thyssen, Professor, MD, DMSc, Principal Investigator — Department of Dermatology and Allergy, Gentofte Hospital, Denmark
Locations (1):
- Department of Dermatology and Allergy, Hellerup, Capital Region, Denmark

REFERENCES:
- [Derived] Gether L, Storgaard H, Kezic S, Jakasa I, Hartmann B, Skov-Jeppesen K, Holst JJ, Pedersen AJ, Forman J, van Hall G, Sorensen OE, Skov L, Ropke MA, Knop FK, Thyssen JP. Effects of topical corticosteroid versus tacrolimus on insulin sensitivity and bone homeostasis in adults with atopic dermatitis-A randomized controlled study. Allergy. 2023 Jul;78(7):1964-1979. doi: 10.1111/all.15690. Epub 2023 Mar 21. PMID 36824052